CLINICAL TRIAL: NCT00600587
Title: Phase Ⅱ Study of Induction Erlotinib Therapy in Stage III A(N2) Non-small Cell Lung Cancer Proceeding to Mediastinoscopy/PET and Thoracotomy/Radiotherapy
Brief Title: Induction Erlotinib Therapy in Stage III A (N2) Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Wen-zhao ZHONG, Guangdong General Hospital, Guangdong Provincial People's Hospital
Organization: GuangdongPPH (Unknown)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CSLC-0702; tarceva-123456-1
Record Dates: First submitted 2008-01-14; First posted 2008-01-25 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Carcinoma, Non-Small-Cell Lung; Genes, erbB-1; tyrosine kinase inhibitor; Neoadjuvant Therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Erlotinib targeted NSCLC population based on EGFR gene analysis(EGFR gene status: activating mutation)
  Interventions: Drug: neoadjuvant erlotinib therapy
- B (Active Comparator): Non-erlotinib targeted NSCLC population based on EGFR gene analysis
  Interventions: Drug: neoadjuvant gemcitabine/carboplatin therapy

INTERVENTIONS:
Drug: neoadjuvant erlotinib therapy — 150mg erlotinib taken once daily and continued uninterrupted for 42 days before evaluation/thoracotomy/radiotherapy.
  Other Names: tarceva
  Arms: A
Drug: neoadjuvant gemcitabine/carboplatin therapy — 3 cycles of neoadjuvant gemcitabine(1250mg/m2,d1,d8)/carboplatin(AUC=5,day1) chemotherapy before evaluation/thoracotomy/radiotherapy.
  Other Names: gemzar
  Arms: B

SUMMARY:
The purpose of this study is to evaluate the value of induction Erlotinib therapy before thoracotomy or radiotherapy in ⅢA-N2 (confirmed by mediastinoscopy or PET) non-small cell lung cancer (NSCLC) selected by epidermal growth factor receptor (EGFR) gene analysis and initial to explore a new treatment strategy for ⅢA-N2 NSCLC.

DETAILED DESCRIPTION:
Stage IIIA non-small-cell lung cancer (NSCLC) is seen in a relatively heterogeneous group of patients with ipsilateral mediastinal (N2) lymph node involvement. The relative roles of different treatment modalities are not clear. Epidermal growth factor receptor (EGFR) tyrosine kinase inhibitors (TKIs) may result in dramatic responses in patients with pulmonary adenocarcinoma carrying EGFR activating mutations. In case reports, the efficacy of perioperative EGFR-TKI therapy in patients with locally advanced NSCLC harboring EGFR gene mutations was satisfactory. Although no prospective data support the use of EGFR-TKIs as induction therapy in stage IIIA-N2 NSCLC, their low toxicity profile and the possibility of a rapid tumor response suggests that prospective trials are required. Therefore, this study evaluated the value of induction erlotinib therapy in IIIA-N2 NSCLC selected by EGFR gene analysis and explored a new treatment strategy for this subset. Erlotinib specifically targets the EGFR TK domain, which is highly expressed and occasionally mutated in various forms of cancer. It binds in a reversible fashion to the adenosine triphosphate (ATP) binding site of the receptor.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Histological or cytological documented
* Resectable NSCLC of stage IIIA-N2 confirmed by mediastinoscopy or PET
* Naive therapy NSCLC
* Candidates should be tolerated with induction therapy and thoracotomy with ECOG performance status 0-2, adequate haematological and Hepatic- renal function and qualified lung function
* Enough tissue samples to perform gene analysis

Exclusion Criteria:

* Small cell lung cancer
* Pregnant or breast-feeding women
* Any unstable systemic disease
* Patients with exposure to investigational drug therapy or other concurrent anticancer therapy outside of this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Response to Neoadjuvant Erlotinib Therapy | a week after completion of the induction erlotinib therapy

SECONDARY OUTCOMES:
disease free survival | every 3 months
overall survival | every 3 months
complete resection rate | 7 days after thoractomy
Toxicity of Neoadjuvant Erlotinib Therapy and postoperative complications | one months after thoractomy

CONTACTS AND LOCATIONS:
Overall Officials: Yi-long WU, MD, Principal Investigator — Guangdong Lung Cancer Institute, Guangdong Lung Cancer Institute, Guangdong Academy of Medical Sciences; Xue-ning YANG, MD, Study Chair — Guangdong Lung Cancer Institute, Guangdong Lung Cancer Institute, Guangdong Academy of Medical Sciences; Wen-zhao ZHONG, MD, Study Director — Guangdong Lung Cancer Institute, Guangdong Lung Cancer Institute, Guangdong Academy of Medical Sciences
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Wu YL, Zhong WZ, Li LY, Zhang XT, Zhang L, Zhou CC, Liu W, Jiang B, Mu XL, Lin JY, Zhou Q, Xu CR, Wang Z, Zhang GC, Mok T. Epidermal growth factor receptor mutations and their correlation with gefitinib therapy in patients with non-small cell lung cancer: a meta-analysis based on updated individual patient data from six medical centers in mainland China. J Thorac Oncol. 2007 May;2(5):430-9. doi: 10.1097/01.JTO.0000268677.87496.4c. PMID 17473659
- [Background] Costa DB, Kobayashi S, Tenen DG, Huberman MS. Pooled analysis of the prospective trials of gefitinib monotherapy for EGFR-mutant non-small cell lung cancers. Lung Cancer. 2007 Oct;58(1):95-103. doi: 10.1016/j.lungcan.2007.05.017. Epub 2007 Jul 3. PMID 17610986
- [Background] Takamochi K, Suzuki K, Sugimura H, Funai K, Mori H, Bashar AH, Kazui T. Surgical resection after gefitinib treatment in patients with lung adenocarcinoma harboring epidermal growth factor receptor gene mutation. Lung Cancer. 2007 Oct;58(1):149-55. doi: 10.1016/j.lungcan.2007.04.016. Epub 2007 Jun 4. PMID 17548126
- [Background] Kappers I, Klomp HM, Burgers JA, Van Zandwijk N, Haas RL, van Pel R. Neoadjuvant (induction) erlotinib response in stage IIIA non-small-cell lung cancer. J Clin Oncol. 2008 Sep 1;26(25):4205-7. doi: 10.1200/JCO.2008.16.3709. No abstract available. PMID 18757336
- [Background] Mok TS, Wu YL, Thongprasert S, Yang CH, Chu DT, Saijo N, Sunpaweravong P, Han B, Margono B, Ichinose Y, Nishiwaki Y, Ohe Y, Yang JJ, Chewaskulyong B, Jiang H, Duffield EL, Watkins CL, Armour AA, Fukuoka M. Gefitinib or carboplatin-paclitaxel in pulmonary adenocarcinoma. N Engl J Med. 2009 Sep 3;361(10):947-57. doi: 10.1056/NEJMoa0810699. Epub 2009 Aug 19. PMID 19692680
- [Background] Robinson LA, Wagner H Jr, Ruckdeschel JC; American College of Chest Physicians. Treatment of stage IIIA non-small cell lung cancer. Chest. 2003 Jan;123(1 Suppl):202S-220S. doi: 10.1378/chest.123.1_suppl.202s. PMID 12527580
- [Derived] Zhong W, Yang X, Yan H, Zhang X, Su J, Chen Z, Liao R, Nie Q, Dong S, Zhou Q, Yang J, Tu H, Wu YL. Phase II study of biomarker-guided neoadjuvant treatment strategy for IIIA-N2 non-small cell lung cancer based on epidermal growth factor receptor mutation status. J Hematol Oncol. 2015 May 17;8:54. doi: 10.1186/s13045-015-0151-3. PMID 25981169